CLINICAL TRIAL: NCT02464267
Title: Developing and Validating a Patient-reported Outcome Instrument to Monitor Symptom Management in Pulmonary Exacerbation of Patients Living With Cystic Fibrosis - Item Development
Brief Title: Developing and Validating a Patient-reported Outcome Instrument to Monitor Symptom Management in Pulmonary Exacerbation in CF
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZK-Nr. 2014-0712
Record Dates: First submitted 2015-04-22; First posted 2015-06-08 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis
Keywords: patient reported outcome instrument
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to develop a reliable and valid instrument to measure symptom management (experience and / or management strategies) during exacerbation episodes in CF patients. For the development a sequential exploratory two phase mixed-method study will be applied. In a first step, up to 25 CF patients will be interviewed: approximately 15 CF patients who experienced at least one episode of exacerbation in the past year and approximately CF 10 patients who are currently experiencing an exacerbation. The latter group will be interviewed up to 3 times during and after the antibiotic treatment. The instruments initial item list will be developed on basis of the interviews. Up to five health professionals will rate the items' relevance. In a further step, items' clarity and relevance will be assessed by cognitive debriefing interviews with no more than 10 patients. In the last step (part III), the instrument's preliminary construct and concurrent validity and reliability will be tested in a larger sample up to 150 patients experiencing exacerbation. Patients will be asked to complete the newly developed questionnaires and a set of other questionnaires at one time point. For part III, ethic approval will be asked at a later date (2015).

ELIGIBILITY:
Inclusion Criteria:

Part I A & II:

1. Patients with a confirmed diagnosis of cystic fibrosis
2. Age ≥ 18
3. Experience of at least one exacerbation during the last year requiring antibiotic treatment (oral or intravenous)

Part I B:

1. Patients with a confirmed diagnosis of cystic fibrosis
2. Age ≥ 18
3. Experience of an acute exacerbation requiring antibiotic treatment (oral or intravenous)

Exclusion Criteria:

Part I & II

1. Do not speak or understand German
2. Inability to verbally communicate
3. Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in patient experience of symptom management | Patients will be followed up for 4 weeks after start of antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Schmid-Mohler, Principal Investigator — Centre of Clinical Nursing,
Locations (1):
- University Hospital Zurich, Zurich, Switzerland